CLINICAL TRIAL: NCT00793897
Title: A Phase I Multiple Ascending Dose Study of BMS-754807 in Combination With Paclitaxel and Carboplatin in Subjects With Advanced or Metastatic Solid Tumors
Brief Title: Multiple Dose Study In Cancer Patients: Safety and Tolerability of BMS-754807 in Combination With Paclitaxel and Carboplatin in Patients With Advanced or Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA191-005
Record Dates: First submitted 2008-11-17; First posted 2008-11-19 (Estimated); Last update posted 2012-07-13 (Estimated); Status verified 2012-07

CONDITIONS: Advanced Solid Tumors; Metastatic Solid Tumors
Keywords: Subjects with Advanced or Metastatic Solid Tumors or Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — BMS 754807; Paclitaxel; BMS 181339; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sequential allocation of patients in two dosing schedules (Experimental)
  Interventions: Drug: BMS-754807; Drug: Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: BMS-754807 — Tablets, Oral, escalating doses starting at 10 mg, continuous or intermittent, until disease progression, unacceptable toxicity or at the subject's request
  Other Names: IGF-IR
Drug: Paclitaxel — Vials, IV, 200 mg/m2, Day 1 of a 21-day cycle, until disease progression, unacceptable toxicity or at the subject's request
  Other Names: Taxol; BMS-181339
Drug: Carboplatin — Vials, IV, 6 mg/mL.min, Day 1 of a 21-day cycle, until disease progression, unacceptable toxicity or at the subject's request
  Other Names: Paraplatin; BMY-26575

SUMMARY:
A Phase I dose escalation study to determine the safety, tolerability, pharmacodynamics and preliminary anti-tumor activity of BMS-754807 in combination with chemotherapy drugs, paclitaxel and carboplatin, in patients with advanced or metastatic solid tumors. In addition, the study is expected to identify the recommended dose or dose range of BMS-754807 in combination with paclitaxel and carboplatin for Phase 2 studies

ELIGIBILITY:
Inclusion Criteria:

* Subjects with advanced or metastatic solid tumors for whom carboplatin and paclitaxel is considered an appropriate therapy
* ECOG performance status 0-1
* At least 4 weeks between surgery or last dose prior anti-cancer therapy

Exclusion Criteria:

* Symptomatic brain metastases
* Any disorder or dysregulation of glucose homeostasis {e.g. diabetes)
* Uncontrolled or significant cardiovascular disease
* Inadequate bone marrow, liver or kidney function
* Evidence of > Grade 1 peripheral neuropathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2009-04; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Safety: Toxicities will be evaluated according to the NCI Common Toxicity Criteria for Adverse Events (CTCAE) version 3 | Continuous assessment throughout the duration of the trial: starting with dosing on Day 1 until after 30 day follow-up following the last dose

SECONDARY OUTCOMES:
Pharmacodynamics: Biochemical parameters of drug action in serum | assessed every 6 weeks of the study
Metabolic measures: Effects of the drug on parameters of glucose homeostasis | assessed every 6 weeks of the study
Efficacy Measures: PET scans and tumor assessments by CT/MRI | a total of 3 PET scans at screening and during the first 3 weeks. CT/MRI assessed every 6 weeks
Pharmacokinetic Measures: Blood samples will be collected during pre-specified times | Day 2, 8 and 15 of Cycle 1 and on Day 1 or Cycle 2 (for Arm A subjects only)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (5):
- Australia (2):
  - Local Institution, East Melbourne, Victoria
  - Local Institution, Parville, Victoria
- Canada (2):
  - Local Institution, Edmonton, Alberta
  - Local Institution, Hamilton, Ontario
- Local Institution, Seoul, South Korea

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx